CLINICAL TRIAL: NCT04143100
Title: Anxiety, Symptom Burden, and Dialysis Adherence in In-center Hemodialysis Patients
Brief Title: Anxiety and Symptom Burden in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 19-06020314
Record Dates: First submitted 2019-10-24; First posted 2019-10-29 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Anxiety; ESRD
MeSH Terms: conditions — Anxiety Disorders; Kidney Failure, Chronic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — For our primary analysis (multiple regression) scores on the GAD-7, BAI and PHQ-9 will be used to predict dialysis adherence, as defined as minutes reduced (total dialysis prescribed -total actual time on machine) while controlling for age and gender.

SUMMARY:
Anxiety has been identified as a prevalent and significant co-morbid condition in patients with End Stage Renal Disease (ESRD) being treated with hemodialysis. In particular, anxious sensitivity to symptoms commonly experienced by dialysis patients may lead patients to prematurely terminate their dialysis sessions and may have consequences on their dialysis adequacy and overall quality of life.

The proposed study will examine the relationships between anxiety, depression, quality of life, symptom burden and dialysis prescription adherence. The primary regression analyses will be used to predict the influence of anxiety and depression (independently and together) on measures of adherence behaviors.

DETAILED DESCRIPTION:
Additional analyses will examine the relationship of elevated anxiety and depression scores on symptom burden, QOL, and other measures of dialysis adherence. Retrospective data of the preceding three months will be used to calculate measures of dialysis adherence (shortening and skipping) and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Receiving In-center hemodialysis

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at The Rogosin Institute (Rogosin) hemodialysis treatment facilities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | This is a cross-sectional study, with anxiety scores being correlated with previous 6 months of adherence data
  Anxiety measure - higher scores indicate more anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cukor, PhD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No